CLINICAL TRIAL: NCT00176267
Title: Paclitaxel, Carboplatin And Low Dose Radiation As Induction Therapy In Locally Advanced Head And Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Susanne Arnold (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Susanne Arnold, Associate Director for Clinical Translation, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02-H&N-15-BMS
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Squamous Cell Carcinoma
Keywords: head and neck; squamous cell carcinoma; squamous cell; carcinoma; paclitaxel; carboplatin; radiotherapy; induction therapy
MeSH Terms: conditions — Carcinoma, Squamous Cell; Carcinoma | interventions — Radiotherapy; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Radiation: Radiotherapy; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Radiation: Radiotherapy — 50 cGy on days 1, 2, 8, 15, 22, 23, 29 & 36 of chemotherapy
Drug: Paclitaxel — 75 mg/m2 intravenously over one hour on Days 1, 8, 15, 22, 29 and 36
Drug: Carboplatin — AUC of 6 on Days 1 & 22

SUMMARY:
This study is being performed utilizing two cycles of Paclitaxel and Carboplatin, plus low doses radiation as initial therapy prior to other treatment (surgery or radiation). The study is assessing if utilization of low doses radiation as a chemoenhancer will further increase the response rate seen with initial therapy.

DETAILED DESCRIPTION:
Squamous cell cancers of the head and neck (SCCHN) comprise 5% of all cancers, with 40,000 new cases diagnosed annually. Surgery followed by irradiation or irradiation alone has been the standard of care for locally advanced Stage III and IV patients. With this approach, fewer than 30% of patients achieve long-term remission, and most recur locoregionally. Neoadjuvant chemotherapy has been administered prior to definitive therapy with response rates ranging from 60-90%, with pathologic CR rates documented in 30-70% of clinical responders. However, large randomized trials have shown no improvement in overall survival. Because induction chemotherapy alone does not appear to improve long-term disease free survival in advanced head and neck cancers, concomitant chemotherapy and radiation has been pursued in patients with locally advanced head and neck cancers. The concept of synergy between radiation and chemotherapy is well established in vitro. Various schedules of radiation and chemotherapy have been utilized including weekly chemotherapy during radiation, chemotherapy given every three weeks during radiation and alternating chemotherapy and radiation.

One novel approach to capitalizes on the synergy between radiation and chemotherapy is the use of low doses fractionated radiation (LDFRT) as a chemotherapy enhancer. In vitro data suggests that LDFRT enhances the response of both p53 wild type and p53 mutant cancer cell lines to chemotherapy. Not only was the cell death fraction increased, but there was no development of radioresistance in the cell lines studies when low doses of radiation were utilized. This strategy was translated into a clinical trial using four 80-cGy fractions of radiation with Carboplatin and Paclitaxel. Preliminary results have produced an impressive 85% response rate and this neoadjuvant regimen was safe and easy to deliver in patients with locally advanced SCCHN patients. In recently published work by Belani, a regimen using Carboplatin every four weeks combined with weekly Paclitaxel improved response rates in non-small cell lung cancer. The delivery of chemotherapy on a weekly schedule would be of particular benefit when adding LDFRT, because tumor cells could be exposed to LDFRT on multiple occasions per cycle of induction therapy, without the theoretic development of radioresistance. We propose to expand our understanding of LDFRT and chemotherapy by using two cycles of Paclitaxel and Carboplatin in a modification of the Belani regimen, plus LDFRT as induction therapy prior to definitive treatment (surgery or radiation). It is hoped that using LDFRT as a chemoenhancer will further increase the response rate seen with induction therapy in this population of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients greater than 18 years of age.
2. ECOG performance status of 0, 1 or 2.
3. Patients with pathologically documented bulky T2, III and IV SCCHN (excluding M1 disease), within 2 months of diagnosis. Bulky T2 tumors are defined as those that have a volume of disease greater than 35 cm3 as measured by CT or MRI scan (28).
4. Patients will be medically fit for undergoing chemotherapy. Specifically:

   1. no evidence of active angina pectoris or ventricular arrhythmia's; no myocardial infarction within the last six months. (Patients with medically controlled hypertension or congestive heart failure are eligible.)
   2. an absolute neutrophil count of > 1000/uL and platelet count > 100,000/uL
   3. serum total bilirubin < 1.5 mg/dL
   4. Creatinine Clearance greater than 60 ml/min

      Using an actual or calculated creatinine clearance using the formula:

      (140 - age)x(wgt in kg)*/(serum creatinine)x(72)* multiply by 0.85 for females
   5. if a pre-existing grade I neuropathy exists, patients must be willing to risk worsening neuropathy secondary to Paclitaxel. Patients with grade II or greater neuropathy will be excluded from study.
   6. ability to give written, informed consent to participate in the trial.
5. Patients will have measurable disease as determined by MRI or CT scan or evaluable disease determined by panendoscopy or indirect laryngoscopy to be eligible for enrollment on this study.

Exclusion Criteria:

1. Pregnant females. Males and women of childbearing potential must use effective contraception in order to prevent pregnancy during therapy.
2. Patients with a history of previous or current malignancy at other sites diagnosed within the last 5 years, with the exception of adequately treated carcinoma in-situ of the cervix or basal or squamous cell carcinoma of the skin. Patients with a history of other malignancies, who remain free of recurrence or metastases for greater than five years are eligible.
3. Patients with active infection will not be eligible for this protocol until the infection is treated and the symptoms have clinically resolved.
4. Patients with a history of allergy to drugs utilizing Cremophor in the formulation.
5. Prior chemotherapy, prior irradiation or surgery for SCCHN will not be allowed.
6. Patients with metastatic disease will not be eligible for this study.
7. Patients with grade II or greater peripheral neuropathy will be excluded from study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2002-09; Primary Completion 2005-01 (Actual); Study Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
Response rate | assessed at baseline and once between days 42 and 56, then repeated every 6 months until disease progression
Pathologic complete responses | assessed between 3 and 24 hours after the last dose of radiation

SECONDARY OUTCOMES:
Toxicity | assessed starting day 1 through study completion day 56 or until toxicities resolve
Quality of Life | assessed pre-study and once between study days 42 and 56
Overall survival | throughout study treatment duration and then every 3 months after study completion

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Arnold, MD, Principal Investigator — University of Kentucky